CLINICAL TRIAL: NCT06535893
Title: Sustainable and Efficient Platform of New Therapeutic Development for Early Breast Cancer (S-FACT)
Brief Title: Sustainable and Efficient Platform Trial of New Therapeutic Development for Early Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nagoya City University (Other)
Collaborators: Japan Clinical Oncology Group (Other)
Responsible Party: Principal Investigator, Kazuki Nozawa, Principal Investigator, Nagoya City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG2205
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JCOG2205-TN (Active Comparator): KEYNOTE-522 regimen: Carboplatin + paclitaxel + pembrolizumab followed by doxorubicin + cyclophosphamide + pembrolizumab
  Interventions: Drug: TN
- JCOG2205-TN-1 (Experimental): Carboplatin + paclitaxel + pembrolizumab followed by niraparib + pembrolizumab
  Interventions: Drug: TN-1

INTERVENTIONS:
Drug: TN — Carboplatin + paclitaxel + pembrolizumab followed by doxorubicin + cyclophosphamide + pembrolizumab
  Arms: JCOG2205-TN
Drug: TN-1 — Carboplatin + paclitaxel + pembrolizumab followed by niraparib + pembrolizumab Niraparib Pembrolizumab AC
  Other Names: KEYNOTE-522 regimen
  Arms: JCOG2205-TN-1

SUMMARY:
Randomized phase II trial targeting early-stage breast cancer (stage II-III) applicable to preoperative chemotherapy (NAC), comparing standard treatment with multiple experimental treatments.

DETAILED DESCRIPTION:
This randomized phase II trial targets early-stage breast cancer (stage II-III) with preoperative chemotherapy (NAC). It compares standard treatment with multiple experimental treatments using an adaptive design, allowing new treatments to be added during or after the trial. Patients are classified by subtype and randomized between standard and experimental treatments.

The trial is flexible, permitting single or combination new drug therapies and incorporating circulating tumor DNA (ctDNA) evaluation for precise efficacy and prognosis prediction.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed invasive breast carcinoma
2. Stage II or III
3. ECOG performance status of 0 or 1
4. Age 18-80

Exclusion Criteria:

1. Continuous systemic administration (oral or intravenous) of steroid drugs or other immunosuppressants.
2. History or complication of interstitial lung disease or pulmonary fibrosis diagnosed by imaging or clinical findings.
3. Infection requiring systemic treatment.
4. Active double cancer (however, the following are not excluded: (1) Completely resected cancers: basal cell carcinoma, squamous cell carcinoma at clinical stage I, carcinoma in situ, mucosal carcinoma, superficial bladder carcinoma, (2) Gastrointestinal cancer that has been curatively resected by ESD or EMR, (3) Other cancers that have not recurred for more than 5 years).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2040-06-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | Baseline to surgery
  pCR is defined as the absence of invasive cancer in the breast and sampled regional lymph nodes.
ctDNA clearance rate | Before Neoadjuvant chemotherapy to surgery
  ctDNA test was performed by Natera

CONTACTS AND LOCATIONS:
Locations (1):
- Nagoya City University, Nagoya, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: No